CLINICAL TRIAL: NCT00208806
Title: Clinical Evaluation of Dilated Cardiomyopathy and Cardiac Resynchronization Therapy for Ventricular Dysfunction in Young Patients With and Without Congenital Heart Disease
Brief Title: Resynchronization Therapy in Young Patients With and Without CHD
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Margaret Strieper, Principal Investigator, Emory University
Other Study IDs: 0418-2004
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Dilated Cardiomyopathy; Pediatric
Keywords: Dilated Cardiomyopathy; Pediatric; Bi-ventricular Pacemaker
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- congenital heart patients with congestive heart failure: 20 effected patients with congestive heart failure patients total 50 patients
  Interventions: Other: congestive heart failure patients

INTERVENTIONS:
Other: congestive heart failure patients — observational echo data on congestive heart failure patients

SUMMARY:
Pacemakers can be attached to one or more than one of the heart chambers. After watching pacemakers work over time, doctors have found that the pacemakers that stimulate only one chamber of the heart sometimes lead to problems later. These problems may be changes in the size and shape of the heart. The heart cannot work as well when some of these changes happen. We need to learn more about these changes and how to prevent them. There has not been an easy way to do this. A new treatment called Cardiac Resynchronization Therapy (CRT) is associated with biventricular pacing where two chambers of the heart are stimulated simultaneously. Tissue Doppler Imaging,Tissue Synchronization Imaging and 3 dimensional echocardiography are new forms of technology that look at the heart while it works. They are similar to a moving x-ray that can watch the heart muscles moving. The movement can be measured. Doctors will check for changes that happen over time. This has not been studied in children before because this kind of is new to this group of patients. This technology is noninvasive which means it can be done from the outside of the body and is painless.

The hearts of children grow fast. It is important to be able to know if the pacemaker or problems from dilated cardiomyopathy are causing any changes in the heart that might cause problems. We expect to be able to use information we learn from this study to improve how we use pacemakers in the future to avoid problems that can happen over time.

DETAILED DESCRIPTION:
Hypothesis H1: Children with DCM. Ventricular dyssynchrony is seen in a majority (over 50%) of pediatric patients with DCM.

Specific aim, SA 1: To describe changes in right and left ventricular function using Tissue Synchronization Imaging (TSI),Tissue Doppler Imaging (TDI), 3D echocardiography and conventional echocardiogram parameters in children with dilated cardiomyopathy.

Hypothesis H2: In the pediatric population, clinical signs and symptoms related to dilated cardiomyopathy are improved with the use of biventricular pacing.

Specific aim, SA 2: To quantitate the effects of biventricular pacing therapy on ventricular function in children with dilated cardiomyopathy using Tissue Synchronization Imaging (TSI),Tissue Doppler Imaging (TDI, 3D echocardiography and conventional echocardiographic parameters.

Research Design and Methods

Patient population

The patient population will include children (newborn to 18 years of age) treated for dilated cardiomyopathy at Children's Healthcare of Atlanta (Egleston Campus). Patients receiving pacemaker therapy and medicinal therapy for DCM will be included. For the purpose of this study, dilated cardiomyopathy is defined as an ejection fraction (EF) of <35% with left ventricular (LV) dimensions greater that 95% for age. Only patients with normal heart anatomy and those with repaired congenital defects that have 4 chambers will be evaluated. Heart transplant patients and patients who cannot travel to Children's Healthcare of Atlanta at Egleston for follow-up are excluded from this study. Two distinct patient groups will be examined:

Group 1: Patients with the diagnosis of dilated cardiomyopathy. We will divide these patients into two subgroups:

A: New onset DCM patients (defined as patients who have been diagnosed with DCM within the past 90 days)

B: Established DCM patients (defined as patients who have been diagnosed with DCM for more than 90 days)

Group 2: Paced Patients: Patients with a secondary diagnosis of dilated cardiomyopathy due to chronic RV pacing who are being evaluated for Biventricular pacemaker implantation. This group will also include patients with DCM who have received biventricular pacemakers within the last two years.

The proposed study will be a single center, prospective, pilot evaluation of the ventricular effects of DCM and the effect of Biventricular pacing for the treatment of DCM in pediatric patients. All patients will be enrolled following referral 1) for implantation of a biventricular pacemaker for the treatment of cardiomyopathy or 2) for a research echocardiogram due to the diagnosis of dilated cardiomyopathy without pacemaker therapy. Inclusion criteria will be those children with dilated cardiomyopathy or children referred for biventricular pacemaker implantation or upgrade with the diagnosis of dilated cardiomyopathy. All participants will be required to sign an informed consent prior to any procedures. We anticipate enrolling 50 patients between March 1, 2005 and February 28, 2006 for this study: 25 patients in Group 1 and 25 patients in Group 2. This will give us a confidence level of 95% with a confidence interval of 4-6.

Procedures

Echocardiographic assessment Standard 2-dimensional, M-mode, and Doppler evaluation will be performed. We will assess cardiac function using left ventricular shortening (SF) and ejection fractions (EF measured by Simpson's Rule). We will also perform tissue synchronization imaging (TSI), tissue Doppler imaging (TDI), and 3D echocardiography using the GE Vivid 7 and HP echocardiographic systems. These systems will assist investigators in determining ventricular function and synchrony.

In all, study participants will receive echocardiographic assessment at the following time points:

Group 1 (new onset and established DCM patients without pacemakers):

A) Outpatient with the diagnosis of DCM (no pacemaker)-one echo will be performed at baseline/enrollment;

B) Inpatient with the diagnosis of DCM (no pacemaker)-one echo will be performed within 24 hours of admission to the hospital, 14 days after admission or at discharge from the hospital (whichever comes first), and 3 months 2 weeks after discharge from the hospital.

Group 2 (DCM patients with pacemakers): One echo will be performed at baseline prior to biventricular pacemaker implantation, 14 days after admission or at discharge from the hospital (whichever comes first) following biventricular pacemaker implantation, 2 weeks, 1 month, 3 months, 6 months, 9 months and 12 months 2 weeks after biventricular pacemaker implantation.

Inter-observer variability for each echocardiographic assessment (methods and data analysis) will be performed by Drs. Derek Fyfe and Tracy Froehlich in Non-invasive Cardiology.

Clinical assessment Clinical evaluation, including the collection of concomitant medication administration, number of hospitalizations for heart failure and adverse events will be performed at each visit. An electrocardiogram (EKG) will be performed at all study visits to assess QRS duration. Heart failure functional class will also be collected at every visit using the Ross or NYHA classification.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with dilated cardiomyopathy
* normal heart anatomy or those with repaired congenital defects that have a 4 chambered heart
* referred for a Biventricular pacemaker implantation or upgrade with the diagnosis of dilated cardiomyopathy or for an echocardiogram due to the diagnosis of dilated cardiomyopathy without pacemaker
* signed informed consent

Exclusion Criteria:

* cannot travel back to Children's Healthcare of Atlanta for follow-up
* Patients with a transplanted heart
* no informed consent

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50
Dates: Start 2004-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Strieper, DO, Principal Investigator — Emory University and Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Background] Gras D, Leclercq C, Tang AS, Bucknall C, Luttikhuis HO, Kirstein-Pedersen A. Cardiac resynchronization therapy in advanced heart failure the multicenter InSync clinical study. Eur J Heart Fail. 2002 Jun;4(3):311-20. doi: 10.1016/s1388-9842(02)00018-1. PMID 12034157
- [Background] Cazeau S, Leclercq C, Lavergne T, Walker S, Varma C, Linde C, Garrigue S, Kappenberger L, Haywood GA, Santini M, Bailleul C, Daubert JC; Multisite Stimulation in Cardiomyopathies (MUSTIC) Study Investigators. Effects of multisite biventricular pacing in patients with heart failure and intraventricular conduction delay. N Engl J Med. 2001 Mar 22;344(12):873-80. doi: 10.1056/NEJM200103223441202. PMID 11259720
- [Background] Abraham WT, Fisher WG, Smith AL, Delurgio DB, Leon AR, Loh E, Kocovic DZ, Packer M, Clavell AL, Hayes DL, Ellestad M, Trupp RJ, Underwood J, Pickering F, Truex C, McAtee P, Messenger J; MIRACLE Study Group. Multicenter InSync Randomized Clinical Evaluation. Cardiac resynchronization in chronic heart failure. N Engl J Med. 2002 Jun 13;346(24):1845-53. doi: 10.1056/NEJMoa013168. PMID 12063368
- [Background] Janousek J, Vojtovic P, Hucin B, Tlaskal T, Gebauer RA, Gebauer R, Matejka T, Marek J, Reich O. Resynchronization pacing is a useful adjunct to the management of acute heart failure after surgery for congenital heart defects. Am J Cardiol. 2001 Jul 15;88(2):145-52. doi: 10.1016/s0002-9149(01)01609-5. PMID 11448411
- [Background] Zimmerman FJ, Starr JP, Koenig PR, Smith P, Hijazi ZM, Bacha EA. Acute hemodynamic benefit of multisite ventricular pacing after congenital heart surgery. Ann Thorac Surg. 2003 Jun;75(6):1775-80. doi: 10.1016/s0003-4975(03)00175-9. PMID 12822614